CLINICAL TRIAL: NCT03347006
Title: Exploratory Double Blind Placebo Controlled Study Investigating the Regulation of Proresolving Mediators and White Blood Cell Responses by Fish Oil Supplements in Healthy Volunteers
Brief Title: SPM Regulation by Fish Oil Supplements in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Metagenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 011549; 16/LO/2182 (Other: Research ethics council)
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: SPM Active is the supplement tested in this study
Who Masked: Participant, Investigator
Masking Description: Double blind placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo control
  Interventions: Dietary Supplement: SPM Active
- Dose 1 (Experimental): 1.5 g of omega-3 supplement
  Interventions: Dietary Supplement: SPM Active
- Dose 2 (Experimental): 3.0 g of omega-3 supplement
  Interventions: Dietary Supplement: SPM Active
- Dose 3 (Experimental): 4.5 g of omega-3 supplement
  Interventions: Dietary Supplement: SPM Active

INTERVENTIONS:
Dietary Supplement: SPM Active — Supplement or placebo will be administered orally between 9 am to 9:30 am.
  * Each participant will give a baseline blood sample then they will be given one of the randomly allocated three doses of fish oil supplement, or a matching placebo in one of 8 study groups [this will be on a 1:1:1:1:1:1:1:1 ratio]. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation/placebo, 12ml per time interval.

SUMMARY:
A randomised, double-blind, placebo-controlled study to determine whether fish oil supplementation regulates peripheral levels of specialized pro-resolving mediators and white blood cell responses in healthy volunteers

DETAILED DESCRIPTION:
Rationale for the study The relationship between omega-3 essential fatty acid supplementation, and specifically fish oil supplementation, and SPM production in humans is very poorly understood. Given that the body produces SPM from omega-3 essential fatty acids to regulate inflammation and also to repair damaged tissues, it is critical to gain further insights on how the body utilizes dietary supplementation of omega-3 fatty acids from fish oils for SPM formation. With the availability of a mass spectrometry based platform developed by the investigators the scientific community is now in a unique position to better understand the biology of fish oil supplementation by monitoring the levels of SPM in plasma. This understanding may in turn shed light into the beneficial actions of omega-3 supplementation. It may also provide new leads for the control of excessive inflammation, as found in chronic inflammatory disorders, via dietary supplementation to exploit the body's own defense systems.

Rationale for choice of doses Given that in a study using a different fish oil source and formulation the investigators found that 1 g of essential fatty acids gave a mild but significant increase in plasma SPM levels (25) the investigators chose the lowest dose in the study to be of 1.5g. with the other two doses being within the European Food Safety Authority's Tolerable Upper Intake Level for supplements containing both EPA and DHA. Given that this limit is of 5 g and previous study with both healthy volunteers and patients demonstrated that doses up to 4 g are well tolerated (22-24), the investigators chose the remaining 2 doses to be 3.0 g and 4.5 g. In addition, this supplement was awarded a Generally Recognized as Safe Status (see appendix 1) in the for a dose of up to 5 g. Similar doses of the emulsion from of the fish oil supplement are also being used in an ongoing clinical study in the USA (ClinicalTrials.gov Identifier: NCT02719665) measuring different outcomes to those being investigated in the present study.

Aim of research The aim of this research is to investigate whether fish oil supplementation increases the peripheral blood levels of SPM and whether fish oil supplementation also regulates peripheral white blood cell responses (including neutrophils, monocytes and platelets) to inflammatory stimuli.

Original hypothesis Given that fish oils are rich in omega-3 essential fatty acids that are precursors in the biosynthesis of SPM the hypothesis underlying the present study is: Fish oil supplementation increase peripheral blood levels of SPM precursors that may be converted to bioactive mediators which in turn will regulate white blood cell responses.

ELIGIBILITY:
Inclusion Criteria:

* For participants to be included in the study they will need to meet the following criteria:

  1. Able to provide informed consent
  2. Men and women between the age of 18 and 45
  3. Declare not to be taking aspirin, other NSAIDS, other form of medication or omega-3 fatty acid supplements for more than 2 weeks prior to screening and the duration of the participation.
  4. Willingness to abstain from eating fish for 2 days before each study visit
  5. Willingness to abstain from alcohol consumption for at least 24h prior to each study visit
  6. Willingness to abstain from caffeine as directed before and during study

Exclusion Criteria:

* 1) History of, chronic disorders, cardiovascular disease (e.g., heart disease, stroke), cancer, or diabetes or significant genetically inherited conditions.

  2) Pregnancy or breast-feeding. 3) Hypothyroidism in the opinion of the investigator. 4) Liver disease in the opinion of the investigator. 5) Any abnormality or pre-existing disease which, in the opinion of the investigator, might either expose the subject to risk, or influence the validity of the results.

  6) Women of childbearing potential not taking adequate methods of contraception 7) Inability to read and write in English 8) Participation in a clinical study of a new chemical entity, biological product or a prescription medicine, or loss of more than 400 mL blood, within the previous 3 months 9) Anyone who is currently smoking or used to smoke 10) Presence or history of drug or alcohol abuse or intake of more than the amount of alcohol in the current guidelines on alcohol consumption

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Souza PR, Marques RM, Gomez EA, Colas RA, De Matteis R, Zak A, Patel M, Collier DJ, Dalli J. Enriched Marine Oil Supplements Increase Peripheral Blood Specialized Pro-Resolving Mediators Concentrations and Reprogram Host Immune Responses: A Randomized Double-Blind Placebo-Controlled Study. Circ Res. 2020 Jan 3;126(1):75-90. doi: 10.1161/CIRCRESAHA.119.315506. Epub 2019 Dec 12. PMID 31829100

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Participants will be assigned randomly to this group. They give a baseline blood sample then they will be administered a placebo. Blood will be collected again at 2h, 4h, 6h and 24h after placebo administration, 12ml per time interval. After a minimum interval of 48 hours from the last blood draw, participants will give blood, they will be administered 1.5g of supplement and blood collected at 2h, 4h, 6h and 24h after supplementation, 12ml per time interval. Participants will be asked to return after a minimum of 48 hours from the last blood draw and blood (baseline) will be collected. The participants will be administered a 3 g of marine oils and blood collected after 2h, 4h, 6h and 24h, 12ml per time interval. After a minimum of 48h from the last blood draw participants will donate blood, they will be then given 4.5 g of marine oils and blood drawn 2h, 4h, 6h and 24h after supplementation, 12ml per time interval.
- Group 2: Participants will be assigned randomly to this group. They give a baseline blood sample then they will be administered a 1.5g of marine oils. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation, 12ml per time interval. After a minimum interval of 48 hours from the last blood draw, participants will give blood, they will be administered 3 g of supplement and blood collected at 2h, 4h, 6h and 24h after supplementation, 12ml per time interval. Participants will be asked to return after a minimum of 48 hours from the last blood draw and blood (baseline) will be collected. The participants will be administered a 4.5 g of marine oils and blood collected after 2h, 4h, 6h and 24h, 12ml per time interval. After a minimum of 48h from the last blood draw participants will donate blood, they will be then given placebo and blood drawn 2h, 4h, 6h and 24h, 12ml per time interval.
- Group 3: Participants will be assigned randomly to this group. They give a baseline blood sample then they will be administered a 3 g of marine oils. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation, 12ml per time interval. After a minimum interval of 48 hours from the last blood draw, participants will give blood, they will be administered 4.5 g of supplement and blood collected at 2h, 4h, 6h and 24h after supplementation, 12ml per time interval. Participants will be asked to return after a minimum of 48 hours from the last blood draw and blood (baseline) will be collected. The participants will be administered a placebo and blood collected after 2h, 4h, 6h and 24h, 12ml per time interval. After a minimum of 48h from the last blood draw participants will donate blood, they will be then given 1.5 g of marine oils and blood drawn 2h, 4h, 6h and 24h, 12ml per time interval.
- Group 4: Participants will be assigned randomly to this group. They give a baseline blood sample then they will be administered a 4.5 g of marine oils. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation, 12ml per time interval. After a minimum interval of 48 hours from the last blood draw, participants will give blood, they will be administered placebo and blood collected at 2h, 4h, 6h and 24h later, 12ml per time interval. Participants will be asked to return after a minimum of 48 hours from the last blood draw and blood (baseline) will be collected. The participants will be administered a 1.5 g of marine oils and blood collected after 2h, 4h, 6h and 24h, 12ml per time interval. After a minimum of 48h from the last blood draw participants will donate blood, they will be then given 3 g of marine oils and blood drawn 2h, 4h, 6h and 24h, 12ml per time interval.
- Group 5: Participants will be assigned randomly to this group. They give a baseline blood sample then they will be administered 4.5 g of marine oils. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation, 12ml per time interval. After a minimum interval of 48 hours from the last blood draw, participants will give blood, they will be administered 3g of marine oils and blood collected at 2h, 4h, 6h and 24h later, 12ml per time interval. Participants will be asked to return after a minimum of 48 hours from the last blood draw and blood (baseline) will be collected. The participants will be administered a 1.5 g of marine oils and blood collected after 2h, 4h, 6h and 24h, 12ml per time interval. After a minimum of 48h from the last blood draw participants will donate blood, they will be then given placebo and blood drawn 2h, 4h, 6h and 24h, 12ml per time interval.
- Group 6: Participants will be assigned randomly to this group. They give a baseline blood sample then they will be administered 3 g of marine oils. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation, 12ml per time interval. After a minimum interval of 48 hours from the last blood draw, participants will give blood, they will be administered 1.5 g of marine oils and blood collected at 2h, 4h, 6h and 24h later, 12ml per time interval. Participants will be asked to return after a minimum of 48 hours from the last blood draw and blood (baseline) will be collected. The participants will be administered a placebo and blood collected after 2h, 4h, 6h and 24h, 12ml per time interval. After a minimum of 48h from the last blood draw participants will donate blood, they will be then given 4.5 g of marine oils and blood drawn 2h, 4h, 6h and 24h, 12ml per time interval.
- Group 7: Participants will be assigned randomly to this group. They give a baseline blood sample then they will be administered 1.5 g of marine oils. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation, 12ml per time interval. After a minimum interval of 48 hours from the last blood draw, participants will give blood, they will be administered placebo and blood collected at 2h, 4h, 6h and 24h later, 12ml per time interval. Participants will be asked to return after a minimum of 48 hours from the last blood draw and blood (baseline) will be collected. The participants will be administered a 4.5 g of marine oils and blood collected after 2h, 4h, 6h and 24h, 12ml per time interval. After a minimum of 48h from the last blood draw participants will donate blood, they will be then given 3 g of marine oils and blood drawn 2h, 4h, 6h and 24h, 12ml per time interval.
- Group 8: Participants will be assigned randomly to this group. They give a baseline blood sample then they will be administered placebo. Blood will be collected again at 2h, 4h, 6h and 24h later, 12ml per time interval. After a minimum interval of 48 hours from the last blood draw, participants will give blood, they will be administered 4.5 g of marine oils and blood collected at 2h, 4h, 6h and 24h later, 12ml per time interval. Participants will be asked to return after a minimum of 48 hours from the last blood draw and blood (baseline) will be collected. The participants will be administered a 3 g of marine oils and blood collected after 2h, 4h, 6h and 24h, 12ml per time interval. After a minimum of 48h from the last blood draw participants will donate blood, they will be then given 1.5 g of marine oils and blood drawn 2h, 4h, 6h and 24h, 12ml per time interval.
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8
Started | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 2
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Population: Since this is a crossover study all the participants in this study will recieved all the study interventions ie 1.5g, 3g 4.5g of marine oils and placebo. These will be administered in one of 8 sequences which will be determined by assigning the volunteer to one of 8 study groups.
Arm/Group | Study Population
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants] — Population: This was a cross over study to every participant received each of the treatments
  Participants
    <=18 years | 0
    Between 18 and 65 years | 22
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Study had a cross over design so all participants received all treatments Population: This was a cross over study
  years | 26.41 (4.01)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Study was a cross over study so all participants received all treatments
  Participants
    Female | 13
    Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Study had a cross over design so all participants received all treatments Population: Study had a cross over design so all participants received all treatments
  participants
    United Kingdom | 22
Height [Mean (Standard Deviation); unit: meters] — Study had a cross over design so all participants received all treatments Population: Study had a cross over design so all participants received all treatments
  meters | 1.70 (0.08)
Weight [Mean (Standard Deviation); unit: Kg] — Study had a cross over design so all participants received all treatments Population: Study had a cross over design so all participants received all treatments
  Kg | 68.54 (18.16)
body mass index [Mean (Standard Deviation); unit: kg/m2] — Study had a cross over design so all participants received all treatments Population: Study had a cross over design so all participants received all treatments
  kg/m2 | 23.45 (4.74)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 118.2 (11.39)
Pulse [Mean (Standard Deviation); unit: bpm] | 65.59 (7.64)
Sodium [Mean (Standard Deviation); unit: mmol/L] | 140.4 (2.59)
Potassium [Mean (Standard Deviation); unit: mmol/L] | 4.434 (0.35)
Chloride ions [Mean (Standard Deviation); unit: mmol/L] | 102 (2.00)
Urea [Mean (Standard Deviation); unit: mmol/L] | 4.818 (1.39)
Creatinine [Mean (Standard Deviation); unit: umol/L)] | 79.09 (12.21)
Protein [Mean (Standard Deviation); unit: g/L] | 72.27 (2.83)
Albumin (g/L) [Mean (Standard Deviation); unit: g/L] | 46.59 (2.52)
Bilirubin [Mean (Standard Deviation); unit: µmol/L] | 9.409 (4.93)
adenosine triphosphate [Mean (Standard Deviation); unit: U/L] | 57.5 (11.35)
Alanine aminotransferase [Mean (Standard Deviation); unit: U/L] | 19 (9.20)
Aspartate Transferase [Mean (Standard Deviation); unit: U/L] | 19 (4.22)
Calcium [Mean (Standard Deviation); unit: mml/L] | 2.407 (0.09)
Phosphate (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 1.13 (0.14)
Urate [Mean (Standard Deviation); unit: µmol/L] | 284.3 (59.13)
estimated glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 78.38 (7.87)
Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4.79 (0.79)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 0.929 (0.30)
High density lipoprotein [Mean (Standard Deviation); unit: mmol/L] | 1.765 (0.35)
Low density lipoprotein [Mean (Standard Deviation); unit: mmol/L] | 2.602 (0.75)
Cholesterol -HDL ratio [Mean (Standard Deviation); unit: ratio] | 2.825 (0.68)
non-HDL Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 3.025 (0.84)
White blood cell count [Mean (Standard Deviation); unit: cells*10^6/L] | 6.195 (1.46)
platelet counts [Mean (Standard Deviation); unit: cells 10^9 /L] | 258.6 (60.69)
Hematocrit [Mean (Standard Deviation); unit: L/L] | 0.428 (0.04)
Red blood cell count [Mean (Standard Deviation); unit: cells 10^12/L] | 4.789 (0.42)

OUTCOME MEASURES:

1. Primary Outcome: Increase in the Average Peripheral Blood SPM Levels
Description: The Primary endpoint of the study will be an increase in peripheral blood SPM levels that will be measured calculated by measuring pre-supplement SPM levels to values measured in plasma after supplementation.
Time Frame: outcomes will be measured 24h post supplementation and compared with baseline values (0h)
Population: healthy volunteers
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Placebo: Placebo control
  SPM Active: Supplement or placebo will be administered orally between 9 am to 9:30 am.
  * Each participant will give a baseline blood sample then they will be given one of the randomly allocated three doses of fish oil supplement, or a matching placebo in one of 8 study groups [this will be on a 1:1:1:1:1:1:1:1 ratio]. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation/placebo, 12ml per time interval.
- Dose 1: 1.5 g of omega-3 supplement
  SPM Active: Supplement or placebo will be administered orally between 9 am to 9:30 am.
  * Each participant will give a baseline blood sample then they will be given one of the randomly allocated three doses of fish oil supplement, or a matching placebo in one of 8 study groups [this will be on a 1:1:1:1:1:1:1:1 ratio]. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation/placebo, 12ml per time interval.
- Dose 2: 3.0 g of omega-3 supplement
  SPM Active: Supplement or placebo will be administered orally between 9 am to 9:30 am.
  * Each participant will give a baseline blood sample then they will be given one of the randomly allocated three doses of fish oil supplement, or a matching placebo in one of 8 study groups [this will be on a 1:1:1:1:1:1:1:1 ratio]. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation/placebo, 12ml per time interval.
- Dose 3: 4.5 g of omega-3 supplement
  SPM Active: Supplement or placebo will be administered orally between 9 am to 9:30 am.
  * Each participant will give a baseline blood sample then they will be given one of the randomly allocated three doses of fish oil supplement, or a matching placebo in one of 8 study groups [this will be on a 1:1:1:1:1:1:1:1 ratio]. Blood will be collected again at 2h, 4h, 6h and 24h after supplementation/placebo, 12ml per time interval.
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 22 | 22 | 22 | 22
pg/mL | 56.49 (42.54) | 56.91 (38.50) | 108.8 (110.3) | 139.7 (83.44)

2. Secondary Outcome: Percentage Change in Omega-3 Fatty Acid Levels From Baseline After 24 Hours
Description: Measure ability of peripheral blood neutrophils to uptake S. aureus following pre- and post- supplementation. Looking at relationship between amount of omega-3 fatty acids ingested, the increase in the blood levels of these molecules and white blood cell function.
Time Frame: Outcomes will be measured 24h post supplementation and compared with baseline values (at 0h)
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 22 | 22 | 22 | 22
percent change from baseline | 23.19 (12.90) | 70.01 (28.31) | 22.60 (12.26) | 89.12 (48.61)

3. Secondary Outcome: Changes in the Expression of Peripheral Blood Neutrophil Activation Markers
Description: Changes in the expression of protein linked with neutrophil activation, determined by comparing expression levels of this protein in peripheral blood cells pre- and post supplementation.
Time Frame: outcomes measured 24h post supplementation and compared with baseline values (at 0h)
Measure: Mean (Standard Error); unit: percent change from baseline values
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 22 | 22 | 22 | 22
percent change from baseline values | 31.97 (8.556) | 30.90 (8.379) | 6.723 (5.859) | 13.93 (6.177)

ADVERSE EVENTS:
Time Frame: Up to 1 month after the last supplement/placebo dose was administered, an average of 40 days
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT03347006/Prot_SAP_000.pdf